CLINICAL TRIAL: NCT00355745
Title: Safety and Efficacy of Using CBUS™ System for Ultrasound Breast Imaging Designed for Breast Tumor Diagnosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Helix Medical Systems (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, Helix Medical Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CBUS -RA-001
Record Dates: First submitted 2006-07-22; First posted 2006-07-25 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: Breast; tumor; ultrasound; biopsy; Breast mammographic or ultrasound findings
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

INTERVENTIONS:
Device: Ultrasound breast scanning — breast scanning

SUMMARY:
In the United States, breast cancer is the most common cancer occurring in women (excluding cancers of the skin) and the second most common cause of death from cancer in women (after lung cancer). Approximately 182,800 new cases per year occur in the United States, causing 40,800 death cases per year. Breast cancer is the leading cause of death in women aged 44-50 years. The 5-year survival rate is 60% overall but is greater than 80% for early disease.

If diagnosed at an early stage, breast cancer has an encouraging cure rate: up to 97% of women diagnosed with localized breast cancer will survive five years after their diagnosis. Even if the cancer is found at a more advanced stage, new therapies have enabled many people with breast cancer to experience the same quality of life as before their diagnosis.

Breast ultrasound (US) is an extremely useful modality in the diagnosis of breast disease in the symptomatic clinic. It is routinely used as an adjunct to x-ray mammography and clinical examination and, with younger patients it may be the sole imaging modality. It has well-established value in differentiating between malignant and benign solid lesions in some cases, however, it cannot replace fine needle aspiration and core biopsy.

Conventional breast US scanning is highly operator- dependent, requiring skillful probe manipulation and the mental ability to envisage 3-D tissue structure. Acquiring 3-D US data sets may be advantageous, making it easier to see and interpret 3-D structures, boundaries and interactions.

CBUS™, Circular Breast Ultrasound Scanner is indicated to improve significantly breast images obtained by ultrasound systems. The CBUS™ system automatically acquires a complete breast image and constructs a high quality 3D image of the scanned breast. These images provide diagnostic information of the complete volume of breast tissue including blood flow in a single ultrasonic 3D image.

In this clinical study, the CBUS™ Circular Breast Ultrasound Scanner will be used to automatically image the complete breast and provides a high quality 3D image of the scanned breast.

ELIGIBILITY:
Inclusion Criteria:

* Female age between 21-70 years.
* Subject has mammography or ultrasound findings
* Subject is scheduled for biopsy.
* Subject is scheduled for ultrasound breast scan.
* Subject understands the study procedure.
* Subject is willing to sign the inform consent and comply with the study requirements.

Exclusion Criteria:

* Age < 21 years or > 70 years.
* Subject undergo previous breast surgery
* Known blood coagulation disorders.
* Known cardiac disorders.
* Breast infection / breast abscess / breast pains.
* Ipsilateral breast scar in same quadrant as current lesion
* Recent breast trauma.
* Pregnant or lactating woman
* Subject has bleeding disorder.
* Subject is suffering extreme general weakness.
* Subject objects to the study protocol.
* Physician objection.
* Known cognitive or psychiatric disorder
* Participation in any other clinical trial

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Occurrences of adverse events | immediately

SECONDARY OUTCOMES:
Quality of ultrasound imaging | within 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Levy, PhD, Study Director — Rambam Health Care Campus
Locations (1):
- RAMBAM Medical Center, Haifa, Israel